CLINICAL TRIAL: NCT03767088
Title: Evaluation of Whole-body Electromyostimulation (WB-EMS) in the Context of Inpatient Rehabilitation of Cardiological and Orthopedic Patients by Randomized Controlled Trial
Brief Title: Whole-body Electromyostimulation in Inpatient Rehabilitation
Acronym: GERKO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. Frank Mooren (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Frank Mooren, Prof. Dr. med. (Lehrstuhl für Rehabilitationswissenschaften), University of Witten/Herdecke
Organization: University of Witten/Herdecke (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UWittenHerdecke
Record Dates: First submitted 2018-12-04; First posted 2018-12-06 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Sarcopenia
Keywords: WB-EMS; rehabilitation; sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Intervention Model Description: prospective randomized controlled parallel group design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- WB-EMS (Active Comparator): 1.5 sessions per week; in total: 6 training sessions training duration: 20 min per session stimulation of 8 muscle groups (legs, gluteal region, core, arms) while performing slight eccentric pronounced physiological movement patterns parameters: 85 Hz, 350ms, intermittent, 4 s load vs 4 s regeneration
  Interventions: Device: WB-EMS
- partial WB-EMS (Active Comparator): 1.5 sessions per week; in total: 6 training sessions training duration: 20 min per session stimulation of 2 muscle groups (legs, gluteal region; lower extremities) while performing slight eccentric pronounced physiological movement patterns parameters: 85 Hz, 350ms, intermittent, 4 s load vs 4 s regeneration
  Interventions: Device: WB-EMS
- control (Sham Comparator): active sham comparator: 1.5 sessions per week; in total: 6 training sessions training duration: 20 min per session performing slight eccentric pronounced physiological movement patterns
  Interventions: Other: (synchronized) Training program without WB-EMS

INTERVENTIONS:
Device: WB-EMS — whole body electromyostimulation
  Arms: WB-EMS; partial WB-EMS
Other: (synchronized) Training program without WB-EMS — 20 min of pronounced eccentric movement patterns
  Arms: control

SUMMARY:
Based on various studies, scientific evidence has proven the effectiveness of whole-body electromyostimulation (WB-EMS) on parameters such as increased physiological performance and body composition.

As a pilot project, the aim of the study is to determine the effect of additional WB-EMS as part of the inpatient four-week rehabilitation of sarcopenic subjects.

DETAILED DESCRIPTION:
The loss of muscle mass in the age-associated process (sarcopenia) is a common indication in the field of orthopedic and cardiac rehabilitation, which may also be reinforced by previous immobilization and disuse of the muscles (atrophy of muscle). Sarcopenia is defined as 2 standard deviations of average of the same sex in middle adult life. The present project focuses on the sarcopenia definition of the Foundation for the National Institutes of Health (FNIH). Their limits are < 0.789 (men) and < 0.512 (women) and are calculated by adding the absolute muscle mass of the extremities divided by the body mass index (BMI).

Due to reduced muscle mass and thus limited strength / performance, the implementation of conventional training tools with regard to generate corresponding intensities is no longer possible, or in persons with additional cardiac or orthopedic restrictions heavily limited.

In view of the existing indications, the alternative training technology whole-body electromyostimulation (WB-EMS) is an adequate training tool for the rehabilitation process. The time-saving (max 20 minutes per training session) and effective training method is characterized by low orthopedic and cardiac stress. Thus, WB-EMS combines both relevant aspects of a joint-friendly training with effects on muscle mass and functionality. Through the simultaneous activation of up to 10 muscle regions with corresponding, subjectively decidedly adjustable intensity per muscle group, up to 2,800 cm2 can be addressed. Synchronized to a motion video, the participants perform light physical exercises in parallel to the current pulses.

The aim of the study is, to evaluate the effect of additional WB-EMS during a 4-week period of inpatient rehabilitation, comparing 3 groups:

1. WB-EMS, stimulating 8 muscle groups (legs,arms, core, gluteal region)
2. partial-WB-EMS, just stimulating the lower extremities (legs, gluteal region)
3. control, just performing the functional, mainly eccentric motion pattern without stimulation

ELIGIBILITY:
Inclusion Criteria:

1. skeletal muscle index (SMI) < 0,789 (men); < 0,512 (women)
2. A general state of good health
3. Medically approved unrestricted sports participation as shown by diagnostic performance test
4. Willingness to provide signed informed consent

Exclusion Criteria:

1. Post-coronary artery bypass graft (ACVB) surgery in the last 3 months
2. Condition after pacemaker and defibrillator implantation
3. renal insufficiency from stage 3a
4. epilepsy
5. feverish diseases or infectious diseases
6. Taking medicines the affect muscle metabolism
7. severe neurological disorders
8. Skin injuries in the area of electrodes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
(isometric) muscle strength of arms, legs and trunk (extenstion) | 4 weeks
  isometric strength [Nm] (DIERs Myoline professional, DIERs International GmbH)
muscle function | 4 weeks
  chair rise test [repetitions; n]
muscle function / submaximal performance test | 4 weeks
  6 minute walking test [distance; m]

SECONDARY OUTCOMES:
muscle mass via multifrequency bioimpedance analysis | 4 weeks
  via multifrequency bioimpedance analysis (BIA, Inbody770, Seoul, Korea)
body fat via multifrequency bioimpedance analysis | 4 weeks
  via multifrequency bioimpedance analysis (BIA, Inbody770, Seoul, Korea)
blood-sample: triglycerides | 4 weeks
  blood-sample
blood-sample: high-density lipoprotein (HDL) | 4 weeks
  blood-sample
blood-sample: low-density lipoprotein (LDL) | 4 weeks
  blood-sample
blood-sample: Crea/glomerular filtration rate (GfR) | 4 weeks
  blood-sample
blood-sample: glutamate oxaloacetate transaminase (GOT) | 4 weeks
  blood-sample
blood-sample: glutamic pyruvic transaminase (GPT) | 4 weeks
  blood-sample
blood-sample: gamma-glutamyl transpeptidase (GGT) | 4 weeks
  blood-sample
blood-sample: creatine kinase (CK) | 4 weeks
  blood-sample
blood-sample: myoglobin | 4 weeks
  blood-sample
blood-sample: sodium | 4 weeks
  blood-sample
potassium | 4 weeks
  blood-sample
life quality | 4 weeks
  questionnaire: Short Form 36 Health Survey (SF-36)
self-efficacy | 4 weeks
  questionnaire: Allgemeine Selbstwirksamkeit Kurzskala (ASKU)
activities of daily living | 4 weeks
  questionnaire: Late-Life Function & Disability Instrument (LLFDI)

CONTACTS AND LOCATIONS:
Overall Officials: Frank C Mooren, Prof, Principal Investigator — Department of Rehabilitation Science
Locations (1):
- Klinik Königsfeld der DRV, Ennepetal, North Rhine-Westphalia, Germany